CLINICAL TRIAL: NCT03112330
Title: A Single-center, Non-randomized, Open, Single-arm Confirmatory Clinical Study to Evaluate the Safety and Efficacy of Platelet Rich Plasma Injection for Patients With Atrophic Rhinitis
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Platelet Rich Plasma Injection for Atrophic Rhinitis
Acronym: ARPRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Sung Won Kim, Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMCENT-01
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Atrophic Rhinitis
Keywords: atrophic rhinitis
MeSH Terms: conditions — Rhinitis, Atrophic

STUDY DESIGN:
Intervention Model Description: Platelet Rich Plasma Injection group : 12 patients anticipated Saline spray group : 12 patients anticipated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- platelet rich plasma injection group (Experimental): To evaluate the safety and efficacy of plasma rich platelet injection on inferior turbinate mucosa in patients with atrophic rhinitis
  Interventions: Device: Plasma rich platelet injection; Device: Saline nasal spray

INTERVENTIONS:
Device: Plasma rich platelet injection — Plasma rich platelet injection with 26-gauge needle and 2cc syringe on inferior turbinate mucosa
Device: Saline nasal spray — two puffs of isotonic saline nasal spray twice daily

SUMMARY:
The goal of the suggested research is to develop a treatment option using platelet rich plasma injection for regeneration of atropic nasal mucosa.

Specific aims of the suggested research is to (1) access the effect of platelet rich plasma in the patients with atropic rhinitis . Moreover, we will (2) compare the conservative treatments including saline nasal irrigation or saline nasal spray.

DETAILED DESCRIPTION:
Clinical trials of platelet rich plasma injection for regeneration of atropic nasal mucosa.

* Injection interval and follow-up duration

  * Injection interval 2 weeks (upto total 3 consecutive injection)
  * Follow-up duration: 6 months
* Observation items, clinical assessment items and evaluation method

  * Access the nasal mucosal status using nasal speculum.
  * Access the nasal mucociliary function using saccharin test (primary outcome; once per month).
  * Fill in the nasal symptom scores using Nasal Obstruction Symptom Evaluation(NOSE) Instrument, Sino-Nasal outcome Test 20, and Visual analog scale (secondary outcome; once per month)
* The other atrophic rhinitis patients who did not want to perform platelet rich plasma injection

  * Random allocation to saline nasal irrigation or saline nasal spray group
  * Perform same observation items, clinical assessment items and evaluation method as well as platelet rich plasma injection group

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Complaint of atrophic rhinitis symptoms including nasal crusting, nasal burning sensation, and postnasal drip
* Atrophic rhinitis view on nasal endoscopic finding
* Patients who informed sufficient about other atrophic rhinitis treatment options including Young's operation, lubricants, or saline irrigation, but, want more other active treatment option.

Exclusion Criteria:

* Platelet related disorders
* Low serum platelet (<100,000/㎕)
* Other hematologic disorders
* Septicemia
* Take anticoagulant drugs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The change of mucociliary clearance function using the saccharin test | 2, 4, 8, 12, and 24th week
  The change in saccharin test time of the 2, 4, 8, 12, and 24th week after first treatment

SECONDARY OUTCOMES:
The change of nasal symptoms using the Nasal Obstruction Symptom Evaluation(NOSE) Instrument | 2, 4, 8, 12, and 24th week
  The change in NOSE total scores of the 2, 4, 8, 12, and 24th week after first treatment
The change of nasal symptoms using the Sino-Nasal outcome Test 20 | 2, 4, 8, 12, and 24th week
  The change in Sino-Nasal outcome Test 20 scores of the 2, 4, 8, 12, and 24th week after first treatment
The change of nasal symptoms using the Visual analog scale | 2, 4, 8, 12, and 24th week
  The change in Visual analog scale scores of the 2, 4, 8, 12, and 24th week after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Kim, MD, PhD, Study Chair — Seoul St. Mary's Hospital; Do Hyun Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friji MT, Gopalakrishnan S, Verma SK, Parida PK, Mohapatra DP. New regenerative approach to atrophic rhinitis using autologous lipoaspirate transfer and platelet-rich plasma in five patients: Our Experience. Clin Otolaryngol. 2014 Oct;39(5):289-92. doi: 10.1111/coa.12269. No abstract available. PMID 24938860
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Hildenbrand T, Weber RK, Brehmer D. Rhinitis sicca, dry nose and atrophic rhinitis: a review of the literature. Eur Arch Otorhinolaryngol. 2011 Jan;268(1):17-26. doi: 10.1007/s00405-010-1391-z. Epub 2010 Sep 29. PMID 20878413
- [Background] Mishra A, Kawatra R, Gola M. Interventions for atrophic rhinitis. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008280. doi: 10.1002/14651858.CD008280.pub2. PMID 22336840
- [Background] Jaswal A, Jana AK, Sikder B, Nandi TK, Sadhukhan SK, Das A. Novel treatment of atrophic rhinitis: early results. Eur Arch Otorhinolaryngol. 2008 Oct;265(10):1211-7. doi: 10.1007/s00405-008-0629-5. Epub 2008 Mar 4. PMID 18317788
- [Background] Modrzynski M. Hyaluronic acid gel in the treatment of empty nose syndrome. Am J Rhinol Allergy. 2011 Mar-Apr;25(2):103-6. doi: 10.2500/ajra.2011.25.3577. PMID 21679513
- [Background] Canciani M, Barlocco EG, Mastella G, de Santi MM, Gardi C, Lungarella G. The saccharin method for testing mucociliary function in patients suspected of having primary ciliary dyskinesia. Pediatr Pulmonol. 1988;5(4):210-4. doi: 10.1002/ppul.1950050406. PMID 3237448
- [Background] Stavrakas M, Karkos PD, Markou K, Grigoriadis N. Platelet-rich plasma in otolaryngology. J Laryngol Otol. 2016 Dec;130(12):1098-1102. doi: 10.1017/S0022215116009403. PMID 27938467